CLINICAL TRIAL: NCT07391696
Title: Coffee Intake Biomarker Validation and Association With Respiratory Diseases
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National University of Singapore (Other)
Responsible Party: Principal Investigator, Seow Wei Jie, Assistant Professor, National University of Singapore
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: NUS-IRB-2022-414
Record Dates: First submitted 2025-06-01; First posted 2026-02-06 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2025-06

CONDITIONS: Coffee
MeSH Terms: interventions — Tea

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Coffee Dose-Response Intervention (Experimental): Participants receive sequential dietary interventions with Coffee A, Coffee B/C, and Tea A across 12 weeks, interspersed with washout periods. Biological samples and dietary records are collected throughout.
  Interventions: Dietary Supplement: Coffee A; Dietary Supplement: Coffee B; Dietary Supplement: Tea

INTERVENTIONS:
Dietary Supplement: Coffee A — Week 1: coffee A ≤10 g coffee powder for low dose Week 2: non-coffee consumption (post-consumption kinetics) Week 3: coffee A ≤20 g coffee powder for medium dose Week 4: non-coffee consumption (post-consumption kinetics) Week 5: coffee A ≤40 g coffee powder for high dose Week 6: non-coffee consumption (post-consumption kinetics)
Dietary Supplement: Coffee B — Week 7: coffee B ≤40 g coffee powder for high dose Week 8: non-coffee consumption (post-consumption kinetics)
Dietary Supplement: Tea — Week 9: washout Week 10: tea (control) Week 11: non-coffee consumption (post-consumption kinetics)

SUMMARY:
This proposed project aims to identify and validate biomarkers of coffee exposure in the Singapore population, and assess the association between coffee consumption (via biomarker measurements) and risk of respiratory diseases in a prospective multi-ethnic cohort in Singapore.

Specific Aim 1: To identify and quantify urinary/serum metabolite changes that are associated with coffee consumption in a dose-response intervention study.

ELIGIBILITY:
Inclusion Criteria:

* Regular coffee drinkers aged 21-64 years old, Chinese ethnicity

Exclusion Criteria:

* Healthy individuals who are regular coffee and/or tea drinkers, aged 21-64 years old of Chinese ethnicity with no severe medical conditions and are physically-abled, can participate in the research. However, you cannot participate in or will be released from this study if the following conditions or situations apply to you:

  * Ineligible screening survey which will consist of basic demographic information and questions pertaining to inclusion/exclusion criteria such as age, gender, current medications, chronic illness, etc
  * Dislike drinking coffee and tea
  * Pregnant or breastfeeding
  * Certain medications including Zanaflex, Sirasalud, Ketanest S, Spravato and Ephedrine Sulfate (See full list of medication)
  * Present medical conditions: cancer, cardiometabolic diseases, endocrine diseases, depression, anxiety, caffeine/lactose intolerant, fear of needles and/or blood disorders
  * Recent history of major surgical operations
  * Past or current user of oral/systemic hormone treatment or therapies
  * Taken antibiotics in the last 3 months
  * Taking nutritional supplements (that contains coffee/tea-related compounds naturally found in other plants)
  * Not willing to travel to the University for the study
  * Unable to commit to completing all the sessions in the 10-week intervention study

Ages: 21 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-10-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Urinary and serum metabolite changes associated with coffee consumption | 12week
  Urine and serum samples will undergo a combination of targeted and untargeted metabolomic profiling at the Singapore Phenome Centre located at NTU. Briefly, thawed urine, serum, coffee and tea samples will be analysed directly on the UHPLC-TQ-MS. Secondly, to explore potentially novel biomarkers and/or metabolites related to the consumption of the two types of coffee relevant to Singapore (black coffee and coffee with additives), untargeted metabolomics will be conducted on the urine and serum samples.

CONTACTS AND LOCATIONS:
Locations (1):
- Saw Swee Hock School of Public Health, National University of Singapore, Singapore, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-08-22): https://cdn.clinicaltrials.gov/large-docs/96/NCT07391696/Prot_SAP_000.pdf